CLINICAL TRIAL: NCT06421077
Title: Transcutaneous Auricular Vagus Nerve Stimulation （taVNS）Prevents Postoperative Delirium in Elderly Patients: a Randomized Controlled Study
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation Prevents Postoperative Delirium in Elderly Patients
Acronym: Vnstar
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VNS20240510
Record Dates: First submitted 2024-05-10; First posted 2024-05-20 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-01

CONDITIONS: Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- taVNS with "standard-stimulation parameters" (Active Comparator): with a current stimulation frequency of 25 Hz and a pulse width of 250 μs
  Interventions: Device: transauricular auricular vagus nerve stimulation
- taVNS with "low-stimulation parameters" (Sham Comparator): with a current stimulation frequency of 1 Hz and a pulse width of 250 μs.
  Interventions: Device: transauricular auricular vagus nerve stimulation

INTERVENTIONS:
Device: transauricular auricular vagus nerve stimulation — transauricular auricular vagus nerve stimulation

SUMMARY:
According to the 3D-CAM scale, evaluate the incidence of Postoperative Delirium within 5 days after surgery in elderly patients receiving taVNS.The results are expected to provide evidence of the safety and efficacy of perioperative prophylactic use of taVNS in the clinical application of improving postoperative brain health in elderly patients, as well as theoretical and practical basis for subsequent studies or clinical applications.

DETAILED DESCRIPTION:
This study aims to conduct a prospective, randomized controlled clinical trial on the preventive use of taVNS to improve the incidence of Postoperative Delirium(POD) in elderly patients undergoing anesthesia surgery. The intervention group will receive "standard-stimulation parameters" of taVNS（25HZ，250μs）, while the control group will receive "low-stimulation parameters" of taVNS(1HZ,250μs). The main outcome measure of the study was the incidence of POD within 5 days after surgery. Secondary outcome measures include incidence of new mild and severe postoperative neurocognitive impairment during hospitalization and 90 days, all-cause mortality rate at 90 days, incidence of related adverse events, and length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Age≥65 years
* Expected operation time≥ 2 hours
* Postoperative hospital stay≥ 4 days
* Sign the informed consent form

Exclusion Criteria:

* Neurosurgery or cardiac surgery
* Emergency surgery within 6 hours of admission
* End-stage disease with an expected survival of < 3 months
* Preoperative severe cognitive dysfunction affected perioperative cognitive function assessment
* Severe sinus bradycardia, AVB of degree II and above, pacemaker placement

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1776 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of POD at discharge or within 5 days postoperatively | At discharge or within 5 days postoperatively
  POD assessment was performed using the 3D-CAM scale estimate. Assessed 2 times daily until postoperative day 5 or hospital discharge

SECONDARY OUTCOMES:
Incidence of delayed cognitive recovery during hospitalization | Day 1 before surgery, day 5 after surgery, day 90 after surgery
  The MMSE/MoCA scale were used for evaluation
Incidence of neurocognitive dysfunction at 90 days postoperatively | on the 90 days
  assessed by AMTS scale
Degree of decline in activities of daily living at 90 days postoperatively | on the 90 days
  use the IADL score
All-cause mortality | on the 90 days
Incidence of unplanned ICU or HDU admissions | on the 90 days
Proportion of patients requiring higher levels of care postdischarge, specifically long-term care. | on the 90 days
Length of hospital stay | on the 90 days
Delirium severity | At discharge or within 5 days postoperatively
  Delirium severity was assessed via the 3D-CAM-S scale. 3D-CAM-S scale: The total score is 7, with 0 being normal, 1 being mild delirium, 2 being moderate delirium, and 3-7 being severe delirium

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu Y, Hou X, Wang T, Wang X, Zhang K, Liang F, Jian M, Wang B, Liu H, Wang A, Han R. Transcutaneous auricular vagus nerve stimulation prevents postoperative delirium in elderly patients (VNSTAR): protocol for a multicentre, randomised controlled trial. BMJ Open. 2025 May 30;15(5):e099736. doi: 10.1136/bmjopen-2025-099736. PMID 40447430